CLINICAL TRIAL: NCT02791984
Title: Respiratory Variability in Aortic Blood Velocity Measured by Suprasternal View as an Indicator of Fluid Responsiveness
Acronym: SUPRA-PAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL14-0408
Record Dates: First submitted 2016-05-27; First posted 2016-06-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-05

CONDITIONS: Cardiovascular System
Keywords: Suprasternal; echography; fluid responsiveness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluid challenge with 250 ml of Ringer Lactate (Experimental)
  Interventions: Device: Fluid challenge with 250 ml of Ringer Lactate

INTERVENTIONS:
Device: Fluid challenge with 250 ml of Ringer Lactate — Fluid challenge with 250 ml of Ringer Lactate over less than 2 minutes, intra-venous, help by a syringe of 50 ml.
  Measure of peak velocity before and after the fluid challenge

SUMMARY:
Respiratory changes in aortic blood velocity have been described as an indicator of fluid responsiveness when measured in the left ventricular outflow tract by trans esophageal echography. A threshold value of 12% allowed discrimination between responders and nonresponders with a sensitivity of 100% and a specificity of 89%. The suprasternal window is already used to measure cardiac output. The primary endpoint of this study is to determine the predictive value of the respiratory variability in aortic blood velocity measured by suprasternal view (∆VpicSS) as an indicator of fluid responsiveness. The secondary endpoint is to compare maximum velocity and velocity time integral measured by suprasternal and transthoracic view.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* American Society of Anesthesiologists (ASA) score 1 or 2
* General Anesthesia with mechanical ventilation
* General Surgery

Exclusion Criteria:

* Arrhythmia
* Spontaneous breathing activity
* Significant valvular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Percentage of cardiac flow variability | At day 1(before surgery)
  Percentage of cardiac flow variability between the 2 echographic measures. Echographic measures will be realized a first time before fluid challenge by suprasternal view and a second time after the fluid challenge by suprasternal view.

SECONDARY OUTCOMES:
Comparison of percentage of cardiac flow variability between transthoracic and suprasternal views | At day 1(before surgery)
  Echographic measures will be realized a first time before fluid challenge by transthoracic and by suprasternal view and a second time after the fluid challenge by transthoracic and by suprasternal view.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Devauchelle, MD, Principal Investigator — Hopital de la Croix-Rousse
Locations (1):
- Hopital de la Croix-Rousse, Hospices Civils de Lyon, Lyon, France